CLINICAL TRIAL: NCT02825433
Title: Observing Changes in Ventilation Pattern During Procedural Sedation
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lara Brewer, Assistant Research Professor, University of Utah
Other Study IDs: IRB_00061832
Record Dates: First submitted 2016-06-25; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving procedural sedation: The investigators collected ventilation data for each breath (respiratory rate, tidal volume, and end-tidal CO2) for all patients receiving procedural sedation for endoscopy.
  Interventions: Other: No intervention, only ventilation monitoring

INTERVENTIONS:
Other: No intervention, only ventilation monitoring

SUMMARY:
The ventilation (respiratory rate, tidal volume and end-tidal CO2) was monitored for patients receiving procedural sedation during endoscopy procedures in order to observe what changes commonly occur.

DETAILED DESCRIPTION:
The literature does not currently describe which ventilation changes a clinician should watch for to keep a patient safe during procedural sedation provided by fentanyl and propofol. This observational study aimed to record the breath-by-breath respiratory rate, tidal volume and end-tidal CO2 for each patient during procedural sedation for each endoscopy procedure. Data analysis offline will aim to identify any patterns in ventilation which may precede apnea or blood oxygen desaturation. The patterns in ventilation preceding apnea or blood oxygen saturation will be compared and contrasted with the patterns of ventilation during normal ventilation periods.

ELIGIBILITY:
Inclusion Criteria:

* (i) ASA I, II, or III
* (ii) patients older than eighteen
* (iii) English speaking
* (iv) undergoing a colonoscopy procedure and receiving procedural sedation

Exclusion Criteria:

* (i) inability/refusal of subject to provide informed consent
* (ii) standard colonoscopy exclusion criteria used at the GI lab at the University of Utah
* (iii) patients with severe medical conditions that in the view of the acting physician prohibits participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving procedural sedation for endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | Measured for every breath observed throughout the endoscopy procedure
Tidal volume | Measured for every breath observed throughout the endoscopy procedure
End-tidal CO2 | Measured for every breath observed throughout the endoscopy procedure

IPD SHARING:
Plan to Share IPD: No